CLINICAL TRIAL: NCT03860883
Title: Melanoma Margins Trial-II - A Phase III, Multi-centre Randomised Controlled Trial Investigating 1cm v 2cm Wide Surgical Excision Margins for AJCC Stage II Primary Cutaneous Melanoma (02.18 MelMarT-II)
Brief Title: Melanoma Margins Trial-II: 1cm v 2cm Wide Surgical Excision Margins for AJCC Stage II Primary Cutaneous Melanoma
Acronym: MelMarT-II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Melanoma and Skin Cancer Trials Limited (Other)
Collaborators: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other); Canadian Cancer Trials Group (Network); Cancer Trials Ireland (Network); Zuyderland Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02.18
Record Dates: First submitted 2019-02-07; First posted 2019-03-04 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Cutaneous Melanoma, Stage II
Keywords: Malignant; Melanoma; Cancer; Surgery
MeSH Terms: conditions — Melanoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Wide Local Excision = 1cm Margin) (Experimental): 1cm Wide Local Excision margin + Sentinel Lymph Node Biopsy +/- Reconstruction
  Interventions: Procedure: Wide Local Excision = 1cm Margin
- Arm B (Wide Local Excision = 2cm Margin) (Active Comparator): 2 cm Wide Local Excision margin + Sentinel Lymph Node Biopsy +/- Reconstruction
  Interventions: Procedure: Wide Local Excision = 2cm Margin

INTERVENTIONS:
Procedure: Wide Local Excision = 1cm Margin — A wide local excision involves removing an extra "safety margin" of skin surrounding the original melanoma site, to ensure that any remaining scattered melanoma tumour cells that may have been left behind after the first initial biopsy/surgery are removed.
  Arms: Arm A (Wide Local Excision = 1cm Margin)
Procedure: Wide Local Excision = 2cm Margin — A wide local excision involves removing an extra "safety margin" of skin surrounding the original melanoma site, to ensure that any remaining scattered melanoma tumour cells that may have been left behind after the first initial biopsy/surgery are removed.
  Arms: Arm B (Wide Local Excision = 2cm Margin)

SUMMARY:
Patients with a primary invasive melanoma are recommended to undergo excision of the primary lesion with a wide margin. There is evidence that less radical margins of excision may be just as safe. This is a randomised controlled trial of 1 cm versus 2 cm margin of excision of the primary lesion for adult patients with stage II primary invasive cutaneous melanomas (AJCC 8th edition) to determine differences in disease-free survival. A reduction in margins is expected to improve patient quality of life.

DETAILED DESCRIPTION:
This study will determine whether there is a difference in disease-free survival rates for patients with primary cutaneous melanoma with Breslow thickness > 2mm or 1-2mm with ulceration (pT2b-pT4b, AJCC 8th edition), treated with either a 1cm excision margin or 2cm margin. The study is designed to be able to prove or disprove that there is no difference in risk of the tumour recurring around the scar or anywhere else in the body between the two groups of patients. If the study shows no risk of tumour recurrence then we will also be able to determine how much of an impact the narrower excision has on patients in terms of improved quality of life and reduced side effects from the surgery and melanoma disease. This trial will also evaluate and determine the economic impact of narrower excision margins on the health services and society in general.

ELIGIBILITY:
Inclusion Criteria:

Patients may be included in the study if they meet ALL of the following criteria:

1. 1. Patients must have a Stage II primary invasive cutaneous melanoma (pT2b-pT4b, AJCC 8th edition) with Breslow thickness >1.0mm to 2.0mm; >2.0mm to 4.0mm or >4.0mm with ulceration, or >2.0mm to 4.0mm; or >4.0mm without ulceration (Table 1) as determined by diagnostic biopsy (narrow excision, incision, shave or punch biopsy) and subsequent histopathological analysis.
2. Must have a primary melanoma that is cutaneous (including head, neck, trunk, extremity, scalp, palm or sole).
3. An uninterrupted 2cm margin must be technically feasible around biopsy scar or primary melanoma.
4. 4. Surgical intervention (which refers to the staging -SLNB and WLE as these are both to be done on the same day) must be completed within 120 days of the original diagnosis. Surgical intervention must also be performed within 28 days of randomisation.
5. Patients must be 18 years or older at time of consent.
6. Patient must be able to give informed consent and comply with the treatment protocol and follow up plan.
7. Life expectancy of at least 5 years from the time of diagnosis, not considering the melanoma in question, as determined by the PI.
8. Patients must have an ECOG performance score between 0 and 1 at screening.
9. A survivor of prior cancer is eligible provided that ALL of the following criteria are met and documented:

   * The patient has undergone potentially curative therapy for all prior malignancies,
   * There has been no evidence of recurrence of any prior malignancies for at least FIVE years (with the exception of successfully treated uterine/cervical or non-melanoma skin cancers (SCCs/BCCs) with no evidence of recurrence), and
   * The patient is deemed by their treating physician to be at low risk of recurrence from previous malignancies.

Exclusion Criteria:

Patients will be excluded from the study for ANY of the following reasons:

1. Uncertain diagnosis of melanoma i.e., so-called 'melanocytic lesion of unknown malignant potential'.
2. Patient has already undergone WLE at the site of the primary index lesion.
3. Patient unable or ineligible to undergo staging SLNB of the primary index lesion.
4. Perineural invasion or neurotropic melanoma: Neurotropism or perineural invasion in any type of melanoma is an exclusion. Perineural invasion does not include entrapment of nerves within the main primary tumour mass.
5. Desmoplastic melanoma: with any patient where pathology determines melanoma as PURE desmoplastic (as per WHO definition of >90% desmoplasia), they are not eligible for this study. However melanomas with less than 90% desmoplasia or mixed desmoplastic subtypes are eligible unless there is neurotropism present (perineural invasion).
6. Microsatellitosis (a nest of metastatic tumour cells found to be growing away from the primary tumour) as per AJCC 8th edition definition is an exclusion.
7. Subungual melanoma
8. Patient has already undergone a local flap reconstruction of the defect after excision of the primary and determination of an accurate excision margin is impossible.
9. History of previous or concurrent (i.e. >1 primary melanoma) invasive melanoma.
10. Melanoma located distal to the metacarpophalangeal joint; on the tip of the nose; the eyelids or on the ear; genitalia, perineum or anus; mucous membranes or internal viscera.
11. Physical, clinical, radiographic or pathologic evidence of satellite, in-transit, regional, or distant metastatic melanoma.
12. Patient has undergone surgery on a separate occasion to clear the lymph nodes of the probable draining lymphatic field, including -SLNB, of the index melanoma.
13. Any additional solid tumour or hematologic malignancy during the past 5 years (with exception of non- melanoma skin cancers (T1 skin lesions of squamous cell carcinoma (SCCs), basal cell carcinoma (BCCs)), or uterine/cervical cancer).
14. Melanoma-related operative procedures not corresponding to criteria described in the protocol.
15. Planned adjuvant radiotherapy to the primary melanoma site after wide local excision is not permitted as part of the protocol and any patients given this treatment would be excluded from the study.
16. History of organ transplantation.
17. Oral or parenteral immunosuppressive agents (not topical or inhaled steroids) at enrolment or within 6 months prior to enrolment.

Pregnancy is not a specific exclusion criterion for this trial, though it may not be clinically appropriate to perform a wide excision and SLNB until the pregnancy has been completed, which may exclude the patient due to violation of inclusion criterion 4. We would advise careful counselling of the patient prior to enrolling the patient, which would include a discussion at the treating centre's multidisciplinary team meeting or tumour board. We would strongly advise contacting the central trial office to discuss the case prior to enrolling on the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2998 (Estimated)
Dates: Start 2019-12-17 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival | 0-60 months
  Time from randomisation until the first clinically, histologically or radiologically confirmed recurrence of melanoma at any body site, or death from any cause.

SECONDARY OUTCOMES:
Local Recurrence | Day 0-Trial Completion (max. 120 months)
  Time from randomisation to any clinically, histologically or radiologically confirmed LR of melanoma including satellite lesions and in transit metastases between the primary site and the regional draining lymph nodes or death from any cause.
Distant Disease-Free Survival | Day 0-Trial Completion (max. 120 months)
  Time from randomisation to any clinically, histologically or radiologically confirmed distant recurrence of melanoma or death from any cause
Melanoma-Specific Survival | Day 0-Trial Completion (max. 120 months)
  Time from randomisation to death due to melanoma
Overall Survival | Day 0-Trial Completion (max. 120 months)
  Time from randomisation to death from any cause
Melanoma-specific Quality of Life: FACT-M questionnaire | Baseline, 3, 6, 12 & 24 months
  Measured by FACT-M (Functional Assessment of Cancer Therapy - Melanoma) questionnaire - It consists of two subsections: The FACT-G subsection is a 27-item compilation of general questions divided into four primary QOL domains: Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, and Functional Well-Being. It is considered appropriate for use with patients with any form of cancer. The Melanoma Surgery Subscale evaluates melanoma-specific symptoms such as surgical morbidity and side effects.
Neuropathic Pain: PainDetect questionnaire | Baseline, 3, 6, 12 & 24 months
  Measured by PainDetect questionnaire
Health-related Quality of Life: EQ-5D-5L questionnaire | Baseline, 3, 6, 12 & 24 months
  Measured by EuroQoL EQ-5D-5L questionnaire - This tool contains 5 domains including mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
Surgery Related Adverse Events | Up to 12-months from the date of surgery
  The following surgical-related adverse events will be recorded from the time of surgery to 12-months following surgery (inclusive):
  * wound dehiscence
  * seroma/haematoma
  * haemorrhage
  * infection
  * skin graft failure
  * necrosis of flap used for reconstruction
  * deep venous thrombosis
  * urinary tract infection
  * pneumonia
  * cardiac complications
  * lymphoedema
Health Economic Evaluation | Baseline, 3, 6, 12 & 24 months
  Data collected for economic analysis will be from hospital notes, MBS and PBS data (Australia) and patient reported outcome measures (including an employment questionnaire) at baseline, 3, 6, 12 and 24 months and at melanoma recurrence.
Serious Adverse Events | from randomisation up to 12-months post-surgery
  All Serious Adverse events (SAEs), will be recorded from randomisation until 12 months post the surgical intervention or until the patient withdraws or dies.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Henderson, Study Chair — Peter MacCallum Cancer Centre, Australia; Marc Moncrieff, Study Chair — Norfolk & Norwich University Hospital
Locations (190):
- United States (128):
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic Phoenix, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - The Angeles (Cedars-Sinai Medical Center and its Affiliates), Los Angeles, California
  - UC Irvine Health - Chao Family Comprehensive Cancer Center, Orange, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Orange, California
  - Stanford Cancer Institute, Palo Alto, California
  - Huntington Memorial Hospital, Pasadena, California
  - Stanford Cancer Center South Bay, San Jose, California
  - Kaiser Permanente - Vallejo Medical Center, Vallejo, California
  - Kaiser Permanente - Walnut Creek Medical Center, Walnut Creek, California
  - Smilow Hospital Care Center, Guilford, Guilford, Connecticut
  - Yale University, New Haven, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - University of Miami Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - University of Miami Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - University of Miami Sylvester Cancer Center at Coral Springs, Coral Springs, Florida
  - University of Miami Sylvester Comprehensive Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Sylvester Comprehensive Center at Hollywood, Hollywood, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Lakeland Regional Health Hollis Cancer Center, Lakeland, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Centre, Miami, Florida
  - University of Miami Comprehensive Cancer Center at Kendall, Miami, Florida
  - University of Miami Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Magnolia Campus, Tampa, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital Atlanta, Atlanta, Georgia
  - Northside Hospital Cancer Institute, Atlanta, Georgia
  - Nancy N and JC Lewis Cancer & Research Pavilion St. Joseph's/Candler, Savannah, Georgia
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Northwestern University, Evanston, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Cancer Center Lake Forest Hospital, Lake Forest, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Indiana University - Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - University of Kansas Hospital - Indian Creek Campus, Overland Park, Kansas
  - University of Kansas Hospital- Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky, Lexington, Kentucky
  - MedStar Franklin Square Medical Center, Baltimore, Maryland
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - University of Michigan - Brighton Center for Specialty Care, Brighton, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - West Michigan Cancer Centre, Kalamazoo, Michigan
  - Siteman Cancer Centre, Barnes Jewish West County, Creve Coeur, Missouri
  - University of Kansas Cancer Center, Kansas City, Missouri
  - Cox South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Medicine - Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medicine, Omaha, Nebraska
  - Cooperman Barnabas Medical Center, Livingston, New Jersey
  - Rutgers Cancer Institute of New Jersey, Piscataway, New Jersey
  - Lovelace Medical Centre-Saint Joseph Square, Albuquerque, New Mexico
  - Lovelace Women's Hospital, Albuquerque, New Mexico
  - Northwell Health Imbert Cancer Center, Bay Shore, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - NYU Langone Medical Center (Winthrop Hospital), Mineola, New York
  - Northern Westchester Hospital, Mount Kisco, New York
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - University of Rochester, Rochester, New York
  - Phelps Memorial Hospital Center, Sleepy Hollow, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - State University of New York Upstate Medical Center-Community Campus, Syracuse, New York
  - Wilmont Cancer Institute at Webster, Webster, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - University of North Carolina Hospitals - Hillsborough Campus, Hillsborough, North Carolina
  - Sanford Broadway Medical Centre, Fargo, North Dakota
  - Sanford Roger Maris Cancer Centre, Fargo, North Dakota
  - University Hospitals Avon Health Center, Avon, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - University Hospitals Geauga Medical Center, Chardon, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Centre, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University Hospitals Chagrin Highlands Medical Centre, Orange, Ohio
  - West Chester Hospital (OH394), West Chester, Ohio
  - University Hospitals St. John Medical Center, Westlake, Ohio
  - OUHSC Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Mercy Health Center - Oncology Hematology, Oklahoma City, Oklahoma
  - Kaiser Sunnyside Medical Center, Clackamas, Oregon
  - Kaiser Permanente Northwest - Oncology Clinic, Portland, Oregon
  - St. Luke's University Health Network - Allentown Cancer Center, Allentown, Pennsylvania
  - St Luke's University Health Network, Bethlehem Campus, Bethlehem, Pennsylvania
  - St Luke's University Health Network, Anderson Campus, Easton, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - St Luke's University Health Network Quakertown Campus, Quakertown, Pennsylvania
  - St. Luke's University Health Network - Upper Bucks, Quakertown, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Intermountain Medical Center, Murray, Utah
  - Huntsman Cancer Institute (The University of Utah), Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermount and Sate Agricultural College, Burlington, Vermont
  - University of Virginia Health System, Charlottesville, Virginia
  - VCU Massey Cancer Center Peninsula Cancer Institute, Newport News, Virginia
  - VCU Massey Cancer Center, Richmond, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - VCU Massey Cancer Center Affiliate Valley Health, Winchester, Virginia
  - University of Winsconsin Carbone Cancer Center-Eastpark medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Marshfield Medical Center - Marshfield, Marshfield, Wisconsin
  - Aurora St Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Medical Center- Weston, Weston, Wisconsin
- Australia (10):
  - Calvary Public Hospital Bruce, Bruce, Australian Capital Territory
  - The Canberra Hospital, Garran, Australian Capital Territory
  - Westmead Hospital, Sydney, New South Wales
  - Melanoma Institute Australia, Sydney, New South Wales
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Robina Hospital, Gold Coast, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Canada (12):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - BCCA - Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Hamilton Health Sciences Centre, Hamilton, Ontario
  - Oak Valley Health, Markham, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - UHN - Princess Margaret Cancer Centre, Toronto, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - Hotel-Dieu de Quebec, Québec, Quebec
- Ireland (3):
  - Cork University Hospital, Cork
  - Mater Misericordiae University Hospital, Dublin
  - St James Hospital, Dublin
- Italy (3):
  - IOV Istituto Oncologico Veneto IRCCS-Padova, Padua
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - AOU Città della Salute e della Scienza di Torino, Torino
- Netherlands (10):
  - Flevo Hospital, Almere Stad, Flevoland
  - Ziekenhuis Gelderse Vallei, Ede, Gelderland
  - Gelre Hospital, Zutphen, Gelderland
  - Maxima Medical Centre, Eindhoven, Eindhoven, North Brabant
  - University Medical Centre Groningen, Groningen
  - Zuyderland Medical Center, Heerlen
  - Maastricht University Medical Center, Maastricht
  - Diakonessenhuis, Utrecht
  - Maxima Medical Center - Veldhoven, Veldhoven
  - Isala Hospital, Zwolle
- North Shore Hospital, Auckland, New Zealand
- Institute of Oncology Ljubljana, Ljubljana, Slovenia
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Central Hospital Kristianstad, Kristianstad
- United Kingdom (20):
  - University Hospitals Birmingham NHS Foundation Trust, Edgbaston, Birmingham
  - Royal Cornwall Hospital NHS Trust, Truro, Cornwall
  - Hull University Teaching Hospitals NHS Trust, Hull, East Yorkshire
  - MID & South Essex NHS Foundation Trust, Westcliff-on-Sea, Essex
  - Lancashire Teaching Hospitals NHS Foundation Trust, Preston, Lancashire
  - Oxford University Hospitals NHS Foundation Trust, Headington, Oxford
  - Imperial College Healthcare NHS Trust, London, The Bays
  - Queen Victoria Hospital NHS Foundation Trust, East Grinstead, West Sussex
  - North Bristol NHS Trust, Bristol
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - The Leeds Teaching Hospitals NHS Trust, Leeds
  - St. Helens & Knowsley Teaching Hospitals NHS Trust, Liverpool
  - Royal Free London NHS Foundation Trust, London
  - Guy's and St Thomas's NHS Foundation Trust, of St Thomas' Hospital, London
  - St George's University Hospitals NHS Foundation Trust, London
  - The Royal Marsden Hospital NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - South Tees Hospitals NHS Foundation Trust of The James Cook University Hospital, Middlesbrough
  - Norfolk and Norwich University Hospital NHS Trust, Norwich
  - Nottingham University Hospitals, NHS Trust, Trust HQ, City Hospital, Nottingham

IPD SHARING:
Plan to Share IPD: No